CLINICAL TRIAL: NCT06181461
Title: Effects of Gong's Versus Kaltenborn Mobilization on Pain, Range of Motion and Function in Patients With Adhesive Capsulitis
Brief Title: Gong's Versus Kaltenborn Mobilization on Pain, Range of Motion and Function in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-528-09-2023
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2023-12

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gong's Mobilization (Experimental): Group A received Gong's mobilization with routine physical therapy included a 30-45 min session with 15-min TENS. Patients followed daily care instructions, using the affected shoulder in daily activities, and performed pendulum and active shoulder exercises twice a day.
  Interventions: Other: Gong's Mobilization
- Kaltenborn Mobilization (Experimental): Group B will receive Kaltenborn mobilization (Grade III posterior translation) with routine therapy. Posterior translation is applied in 30-sec sets, repeated 15 times over 10 mins, with 10-sec rests. Routine physical therapy includes 30-45 min sessions with 15-min TENS. Patients follow daily care instructions, use the affected shoulder in daily activities, and perform pendulum and active shoulder exercises twice a day.
  Interventions: Other: Kaltenborn Mobilization

INTERVENTIONS:
Other: Gong's Mobilization — Group A received Gong's mobilization with routine physical therapy included a 30-45 min session with 15-min TENS. Patients followed daily care instructions, using the affected shoulder in daily activities, and performed pendulum and active shoulder exercises twice a day.
  Arms: Gong's Mobilization
Other: Kaltenborn Mobilization — Group B will receive Kaltenborn mobilization (Grade III posterior translation) with routine therapy. Posterior translation is applied in 30-sec sets, repeated 15 times over 10 mins, with 10-sec rests. Routine physical therapy includes 30-45 min sessions with 15-min TENS. Patients follow daily care instructions, use the affected shoulder in daily activities, and perform pendulum and active shoulder exercises twice a day.
  Arms: Kaltenborn Mobilization

SUMMARY:
The study will be a Randomized Clinical Trial set to take place at the Department of Physical Therapy, University of Lahore Teaching Hospital, Defence Road, Lahore. It is projected to span 9 months, beginning after the approval of the synopsis. The calculated sample size, utilizing Visual Analogue Scale as an outcome measure with a 20% dropout consideration, will be 34 in each group. Ethical approval from the Research Ethical Committee will be sought, and participant referrals will be facilitated by orthopedic physicians. Eligibility screening will be carried out, and willing participants will be randomized into Experimental and Comparative groups using a lottery method. The study will maintain single-blinding, with assessors remaining unaware of group allocation.

DETAILED DESCRIPTION:
This research is centered on the comparative effectiveness of Gong's and Kaltenborn's mobilization techniques in the treatment of Adhesive Capsulitis, addressing a significant void in current literature. Prior studies have individually showcased the efficacy of both techniques in enhancing pain relief, expanding range of motion, and improving functional outcomes among patients. However, a direct comparative analysis between Gong's and Kaltenborn's mobilization is conspicuously absent, prompting this study to unveil potential distinctions in their impact on shoulder pain, range of motion, and functional mobility.

The research design involves the random allocation of participants into two groups: Group A, receiving Gong's mobilization, and Group B, undergoing Kaltenborn's mobilization. This allocation will be done through a lottery method, ensuring a fair and unbiased selection process. The study will follow a single-blind design, with the assessor remaining unaware of the treatment group assignment.

Participants in both groups will also receive routine physical therapy, including 15 minutes of electrical muscle stimulation with heat therapy. This approach, supported by existing literature, aims to create a standardized baseline for assessing the additional impact of mobilization techniques. The study's duration is projected to be nine months, with data collection points at baseline, the end of 1.5 weeks, and the conclusion of the 3rd week.

Outcome variables include pain assessment using the Numeric Pain Rating Scale, evaluation of function through the Shoulder Pain & Disability Index, and measurement of range of motion using goniometry. Data collection will be performed by an assessor at specified intervals, allowing for a comprehensive understanding of the interventions' effects over time.

Ultimately, this research aspires to contribute evidence-based insights into the relative effectiveness of Gong's and Kaltenborn's mobilization techniques, aiding clinicians in making informed decisions for optimal patient outcomes in the context of Adhesive Capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40-60 years
* Both Male and females
* Patients diagnosed with idiopathic Adhesive Capsulitis
* Patients with 2nd and 3rd stage of Adhesive Capsulitis
* Having at least 5 score of Numeric Pain Rating Scale

Exclusion Criteria:

* Patients with neurological disorders(Thoracic Outlet Syndrome)
* Patients with musculoskeletal disorder(e.g. Rotator Cuff Injury)
* Recent fracture/dislocation in and around the shoulder

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
The Shoulder Pain & disability Index (SPADI) | 3 weeks
  The Shoulder Pain & Disability Index (SPADI) was designed to evaluate shoulder pain and impairment in an outpatient setting. Comprising 13 items, it assesses two domains: a 5-item pain subscale and an 8-item disability subscale. In contrast to the Visual Analog Scale (VAS), the SPADI utilizes a 0-10 scale, with patients circling the number that best represents their pain or disability level, ranging from 0 for minor pain to 10 for severe pain. The total score is calculated similarly to the VAS version. Patients have the option to deem one item as not applicable in each subscale, and that specific item is excluded from the overall score, offering a comprehensive yet adaptable assessment of shoulder pain and disability.
Numeric Pain Rating Scale | 3 weeks
  The Numeric Pain Rating Scale (NPRS) serves as a segmented numeric alternative to the Visual Analog Scale (VAS), allowing respondents to choose a whole number (0-10 integers) that most accurately represents the intensity of their pain. Typically presented as a horizontal bar or line, the NPRS is a quick and straightforward assessment tool, taking less than a minute to complete. Scores on the NPRS range from 0 to 10 points, with higher scores indicative of more intense pain. This scale is versatile, as it can be administered verbally, making it suitable for telephone assessments, or graphically for self-completion, offering a practical means of gauging pain intensity.
Universal Goniometer | 3 weeks
  The universal goniometer is a crucial tool for assessing shoulder range of motion (ROM). With its protractor-like design, it allows precise measurement of angles in various planes, aiding clinicians in objectively evaluating flexion, extension, abduction, adduction, internal rotation, and external rotation. This device, aligned with joint axes, provides quantitative data for diagnosing conditions, monitoring progress, and guiding treatment plans in orthopedics and rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gull, MSPT MSK*, Principal Investigator — University of Lahore; Hafiza Sana Ashraf, MSPT MSK, Study Director — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Pakistan